CLINICAL TRIAL: NCT05884957
Title: Role of Nitric Oxide in Diabetic Patients With Erectile Dysfunction: Effect of Tadalafil Therapy
Brief Title: Role of Nitric Oxide in Diabetic Patients With Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Mona Hamza
Record Dates: First submitted 2023-05-10; First posted 2023-06-01 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Erectile Dysfunction; Diabetes Mellitus
MeSH Terms: conditions — Erectile Dysfunction; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients Group (Nitric oxide Assesment) (Active Comparator): Assessment of nitric oxide synthase gene polymorphism in diabetic patients with erectile dysfunction in 30 patients
  Interventions: Diagnostic Test: Nitric oxide synthase gene
- Control Group (Placebo Comparator): 10 healthy people without erectile dysfunction
  Interventions: Diagnostic Test: Nitric oxide synthase gene

INTERVENTIONS:
Diagnostic Test: Nitric oxide synthase gene — Biochemical assessment of serum nitric oxide level pre and post 5 mg tadalafil therapy in diabetic patients with erectile dysfunction and in normal healthy controls.

SUMMARY:
Erectile dysfunction (ED) is defined as penile erection that is insufficient and unsustainable for a satisfactory sexual performance.

The etiology of ED is multifactorial including chronic diseases such as hypertension, diabetes mellitus and coronary artery disease However, the main underlying cause is degenerative changes that result in endothelial dysfunction

DETAILED DESCRIPTION:
Diabetes leads to endothelial dysfunction and a pro-inflammatory state, which reduces the usability and activity of nitric oxide (NO). NO is a powerful force for sustaining penile blood flow.

Diabetes is an estab¬lished risk factor for sexual dysfunction in men; a three-fold increased risk of erectile dysfunction (ED) was documented in diabetics compared with non-diabetic men.

In smooth muscles, NO activates guanyl cyclase and increases cyclic guanosine monophosphate (cGMP) concentration. cGMP activates certain intracellular protein kinases that phosphorylate receptor proteins. Activated protein kinases open the potassium channels and increase the influx of potassium and block the influx of calcium by inhibiting calcium channels. This leads to hyperpolarization and relaxation of smooth muscle. Reduced arteriolar resistance leads to sinusoidal spaces filled with blood. These enlarged sinusoids further increase the intracavernosal pressure by blocking the venous return and producing a rigid erection. cGMP is converted to GMP by phosphodiesterase, which is inhibited by phosphodiesterase 5 (PDE-5) inhibitors.

(NO) has vasodilatory properties and balances RhoA/Rho-kinase-mediated vasoconstriction, which is a predominant mediator of the physiologic induction and maintenance of erections.

Evidences show that functional polymorphisms within endothelial NO synthase (eNOS) gene interfere with normal erectile function.

In humans, the eNOS gene is located on chromosome 7q35-36 and consists of 26 exons spanning 21 kilobases (kb). Several polymorphisms of eNOS have been investigated. More frequently, investigated regions of this gene include a variable number of 27 bp tandem repeats in intron 4 (VNTR), G894T (rs1799983) polymorphism in exon 7 and a T-786C (rs2070744) polymorphism in the promoter region

ELIGIBILITY:
Inclusion Criteria:

1. Diabetic patients with ED.
2. Using tadalafil 5mg

Exclusion Criteria:

1. Patients with history of pelvic trauma or major pelvic surgical intervention.
2. Patients with hypogonadism and hyperprolactinemia.
3. Patients with chronic liver disease or cardio vascular system diseases.
4. History of chronic intake of central nervous system, anti-androgen drugs or other drugs as Tramadol.
5. Smokers.
6. Patients with non-vasculogenic Erectile dysfunction

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
ِAssessments of endothelial nitric oxide synthase In diabetes mellitus | 24 hours
  About 2 milliliter of blood will be evacuated into EDTA containing tubes and will be stored at-80c till the time of genetic assay of nitric oxide synthase gene polymorphism using RELP - PCR technique .

SECONDARY OUTCOMES:
Tadalafil 5milligram (tablets) therapy in diabetic patients | 3 months from starting the therapy
  Evaluate the effect of endothelial nitric oxide synthase gene polymorphism on response to 5 milligram of Tadalafil (tablets) therapy in diabetic patients with erectile dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hassan, Assist.Prof., Principal Investigator — Medical Biochemistry Department, Faculty of Medicine, South Valley University
Locations (1):
- Qena Hospital, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Undecided